CLINICAL TRIAL: NCT03429647
Title: Intraoperative Perfusion Patterns of the Sigmoid Colon During Elective Open Abdominal Aortic Aneurysm Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EK 316/12
Record Dates: First submitted 2018-01-26; First posted 2018-02-12 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sigmoid perfusion (Other): Measured by visible light spectroscopy
  Interventions: Diagnostic Test: visible light spectroscopy

INTERVENTIONS:
Diagnostic Test: visible light spectroscopy — Sigmoid perfusion was assessed using visible light spectroscopy

SUMMARY:
Blood supply to the sigmoid colon during open abdominal aortic aneurysm (AAA) repair is at risk. Ischemia of the sigmoid colon after AAA repair is potentially devastative. No reliable measures to prevent it are available and the underlying mechanisms are poorly understood. The aim of this study is to describe intraoperative perfusion patterns of the sigmoid colon during open AAA repair and their potential impact on postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective open AAA repair between 2013 and 2016 were eligible for this study

Exclusion Criteria:

* No informed consent
* emergency cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
saturation in the sigmoid colon | intraoperative day
  Perfusion rate

CONTACTS AND LOCATIONS:
Overall Officials: Jasmin Zeindler, MD, Principal Investigator — University Hospital, Basel, Switzerland